CLINICAL TRIAL: NCT06353958
Title: A Retrospective Phase IIa Study of Intravenous Allogeneic Non-HLA-Matched, Unrelated Donor Stem Cell, MiSaver (Myocardial Infarction Saver), Infusion for Recent Acute Myocardial Infarction
Brief Title: MiSaver® Stem Cell Treatment for Acute Myocardial Infarction
Acronym: MiSaver®
Status: Completed | Type: Observational
Sponsor: Honya Medical Inc (Industry)
Collaborators: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: MiSaver PIIa
Record Dates: First submitted 2024-03-27; First posted 2024-04-09 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low: Low dosage of MiSaver cells at 0.5x10^7 cells/kg
  Interventions: Drug: MiSaver
- Middle: Middle dosage of MiSaver cells at 1.6x10^7 cells/kg
  Interventions: Drug: MiSaver

INTERVENTIONS:
Drug: MiSaver — MiSaver vials was thawed using a thermostat-controlled mini bath, drawn into a 20ml syringe, and diluted with normal saline and intravenous infused following standard operating procedures, consecutively, until reasching the dosage.
  Patients were premedicated with intravenous antihistamines (such as diphenhydramine) and corticosteroids (such as hydrocortisone) 30-60 minutes before the stem cell infusion. Any unused solution was discarded, and the total volume of injected solution was adjusted to accommodate the total daily fluid volume administered.

SUMMARY:
Despite advancements in treatments, cardiovascular diseases, especially acute myocardial infarction (AMI), remain significant health concerns. This study hypothesized that stem cells could improve left ventricular function post-AMI. An open-label trial was initiated to assess the safety and feasibility of intravenous infusion of ABO blood group-matched allogeneic umbilical cord blood stem cells (USC) prefabricated into MiSaver (Myocardial Infarction Saver) in AMI patients.

Primary Endpoint:

The primary endpoint focused on safety and adverse events over a 12-month observational period. Results showed the treatment was well-tolerated with no AEs attributed to the study product.

Secondary Outcomes:

Secondary outcomes evaluated changes in left ventricular ejection fraction (LVEF) from baseline to 12 months post-treatment. A retrospective study compared eligible controls with low and middle dosage groups.

DETAILED DESCRIPTION:
Cardiovascular diseases, particularly acute myocardial infarction (AMI), persist as significant health concerns despite advancements in pharmaceutical and interventional treatments. Herein,investigators hypothesized stem cells could enhance left ventricular functional outcomes in patients recently afflicted by acute myocardial infarction (AMI). To investigate this hypothesis, investigators initiated an open-label, dose-escalating trial to evaluate the safety and feasibility of intravenous infusion of ABO matched allogeneic umbilical cord blood stem cells (USC), prefabricated into our study product MiSaver (Myocardial Infarction Functional Saver), in patients following recent AMI. Participants were enrolled in cohorts of five, each receiving low or middle dosages (0.5x10^7 and 1.6x10^7 cells/kg, respectively), with infusions administered 2-5 days post-AMI onset.

(Study details for low and middle dose please see study NCT04050163)

Retrospective participants meeting similar inclusion criteria of recent AMI and LVEF < 45% were identified from the study site. Twenty eligible participants were selected as controls and compared for analysis with the low and middle dosage groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 and 80 years
* Diagnosed with AMI within 7 days
* Elevated cardiac enzymes (Creatine Kinase-MB or troponin) greater than 2 times the upper limit of normal
* Presence of regional wall motion abnormality
* LVEF ≤ 45% on echocardiography
* Hemodynamically stable
* Not requiring inotropic support
* Systolic blood pressure below 80mm Hg for less than 1 hour
* Resting heart rate above 100 beats/min for less than 1 hour in the past 24 hours
* Peripheral artery oxygen saturation of ≥97%

Exclusion Criteria:

* Pregnancy or breastfeeding
* Positive adventitious infections (such as HIV, hepatitis)
* Need for coronary artery bypass surgery or anticipated further revascularization procedures during the 6-month study period
* Severe aortic or mitral valve narrowing
* Evidence of life-threatening arrhythmia on baseline electrocardiogram (ECG)
* Inability to receive PCI examination or treatment (including New York Heart Association (NYHA) Fc.IV) due to shortness of breath
* Malignant tumor
* Hematopoietic dysplasia
* Other severe organ disease
* Less than 1 year of life expectancy
* Chronic kidney disease with estimated Glomerular Filtration Rate (eGFR)<20 and/or on renal dialysis

Ages: 41 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Control group were retrospectively data retried from the study site, comprising 20 eligible participants meeting similar inclusion criteria for recent AMI and left ventricular ejection fraction (LVEF) < 45% was compared for analysis with the low and middle dosage groups.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Safety and adverse events events | 12 months
  The primary endpoint focused on safety evaluation and is measure with number of adverse events (AEs) over a 12-month observational period.

SECONDARY OUTCOMES:
Efficacy on ventricular ejection fraction (LVEF) improvement | 12 months
  Changes in left ventricular ejection fraction (LVEF) from baseline to 12 months post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided